CLINICAL TRIAL: NCT05055310
Title: Shanghai Mental Health Center
Brief Title: The Mechanism of MicroRNAs Network in Alzheimer's Disease
Acronym: MicroRNAs AD
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 81571298
Record Dates: First submitted 2020-01-08; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer Disease
Keywords: MicroRNAs; Alzheimer's Disease; Validation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal elderly: normal cognitive group
  Interventions: Diagnostic Test: MicRNAs test
- aMCI: amnestic mild cognitive impairment
  Interventions: Diagnostic Test: MicRNAs test
- AD: Alzhiemer's disease
  Interventions: Diagnostic Test: MicRNAs test

INTERVENTIONS:
Diagnostic Test: MicRNAs test — plasma micRNAs concentration

SUMMARY:
MicroRNAs network, such as MicRNA107 et al, regulate the pathology of Alzheimer's disease and the clinical validation in diagnosis AD.

ELIGIBILITY:
Inclusion Criteria:

* NIA-AA MCI due to AD clinical criteria for MCI due to AD
* NIA-AA AD clinical criteria for AD

Exclusion Criteria:

* Other type of dementia

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: age between 60 to 90 years old.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
MicRNAs diagnosis validation for aMCI | 5 years
  MicRNAs concentration in plasma among three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychogeriatrics，Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China